CLINICAL TRIAL: NCT00905489
Title: An Open-label, Multiple Dose, Cross-over Study to Evaluate the Steady-state Pharmacokinetic Parameters of Nevirapine Extended Release Tablets in HIV-1 Infected Children, With an Optional Extension Phase
Brief Title: A Phase I Multiple Dose Pharmacokinetic Study of Nevirapine Extended Release (XR) in HIV-1 Infected Children.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1518; 2008-005855-61 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-05-06; First posted 2009-05-20 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

ARMS (1):
- Nevirapine IR / Nevirapine XR (Experimental): In this pharmaco-kinetic (PK) cross-over design trial, all patients initially receive nevirapine immediate release and then all patients are switched to nevirapine extended release 200 mg, 300 mg or 400 mg QD. After completing the PK phase patients had the option of continuing treatment with nevirapine XR in the Optional Extension Phase (OEP).
  Interventions: Drug: Nevirapine Immediate Release (IR); Drug: Nevirapine Extended Release (XR)

INTERVENTIONS:
Drug: Nevirapine Immediate Release (IR) — 200 mg Tablet or 50 mg / 5 ml oral suspension
  Other Names: Nevirapine IR
Drug: Nevirapine Extended Release (XR) — 200 mg, 300 mg or 400 mg Tablet formulation
  Other Names: Nevirapine XR

SUMMARY:
The primary objective is to establish the pharmacokinetic (PK) profile at steady state of nevirapine XR in HIV infected children from >=3 to <18 years of age. This phase I trial is an open-label, multiple dose, non-randomized and cross-over study. Patients who have completed the last visit of the PK trial (visit 7) can enter into an Optional Extension Phase (OEP) until the Investigational New Drug (IND) is withdrawn; until nevirapine XR becomes approved and is available by prescription in a given country; or, the patient enrolls in a compassionate use program. During this OEP, nevirapine XR safety and efficacy information will be collected.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent of a parent or legal guardian prior to admission. Active assent must be given by the patient if the child and/or adolescent is capable of understanding the provided study information.
2. HIV-1 infected males or females >= 3 and < 18 years old.
3. BSA >= 0.58 m2 for patients using BSA to calculate nevirapine IR dose; or BW >= 12.5 kg for patients using BW to calculate nevirapine IR dose at screening visit.
4. Treated with a nevirapine IR based regimen for at least 18 weeks prior to screening visit (Visit 1); no modifications in the ARV background therapy within the last 2 weeks prior to screening.
5. An HIV VL of <50 copies/mL while receiving nevirapine IR at the last measure of VL documented in the medical record obtained within a period of 5 months prior to screening visit.
6. An HIV VL of <50 copies/mL at screening visit.
7. A stable or not decreasing CD4+ cell count according to the investigator's opinion.
8. Acceptable screening laboratory values that indicate adequate baseline organ function according to the opinion of investigator.
9. ALT and AST <= 2.5 X ULN (DAIDS Grade 1).
10. Serum creatinine levels <= 1.3 X ULN (DAIDS Grade 1).
11. Patients able to swallow tablets.

Exclusion criteria:

1. Any AIDS-related or AIDS defining illness that is unresolved or not stable on treatment at least 8 weeks prior to screening visit.
2. Diseases other than HIV infection or conditions that, in the investigator's opinion, would interfere with the study.
3. Patients who have been diagnosed with malignant disease and who are receiving systemic chemotherapy or are anticipated to receive any therapy during their participation in this trial.
4. Use of investigational medications or vaccines within 28 days prior to Visit 1 or during the trial.
5. Use of immunomodulatory drugs within 28 days before Visit 1 or during the trial (e.g., interferon, cyclosporin, hydroxyurea, interleukin 2).
6. Concomitant protease inhibitor (PI) treatment.
7. Unwillingness to abstain from ingesting substances during the study which may alter plasma drug concentrations by interaction with the cytochrome P450 system (Appendix 10.2).
8. Female patients of childbearing potential who:

   * have a positive serum pregnancy test at screening,
   * are breast feeding,
   * are planning on becoming pregnant,
   * are not willing to use double-barrier methods

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- United States (2):
  - 1100.1518.0001 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1100.1518.0002 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
- Botswana (3):
  - 1100.1518.2605 Boehringer Ingelheim Investigational Site, Francistown
  - 1100.1518.2601 Boehringer Ingelheim Investigational Site, Gaborone
  - 1100.1518.2603 Boehringer Ingelheim Investigational Site, Gaborone
- Germany (3):
  - 1100.1518.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1518.4901 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1100.1518.4903 Boehringer Ingelheim Investigational Site, München
- South Africa (2):
  - 1100.1518.2702 Boehringer Ingelheim Investigational Site, Cape Town
  - 1100.1518.2703 Boehringer Ingelheim Investigational Site, Parow Valley

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter Phase I study in Botswana, Germany, South Africa and the United States.
Pre-assignment Details: There was only one treatment group and no randomization process. Overall, 90 pediatric patients were enrolled. Five patients were not entered and 85 patients entered the study. Patients were stratified to the following three age groups: (26 in the 3 - <6 year age group, 26 in the 6 - < 12 year age group and 33 in the 12 - < 18 year age group).
Groups:
- Total.: All patients enrolled in study.
  All patients initially receive nevirapine immediate release (IR) and then all patients are switched to nevirapine extended release (XR) 100mg or 400mg tablets for a once daily dosing of 200 mg, 300 mg or 400 mg QD. After completing the PK phase patients had the option of continuing treatment with nevirapine XR in the Optional Extension Phase (OEP).
Period: Pharmaco-kinetic (PK) Phase
Arm/Group | Total.
Started | 85
Completed | 80
Not Completed | 5
Not completed — Protocol Violation | 2
Not completed — Other reason not defined above | 3
Period: Optional Extension Phase (OEP)
Arm/Group | Total.
Started | 40 (Includes only subjects who chose to continue trt with nevirapine XR after completing the PK phase.)
Completed | 39
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Total.
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Trough Cpre,N.
Description: Trough Nevirapine concentration immediately prior to the next scheduled dose. Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 22.
  The measure of dispersion presented is the coefficient of variation (%) rather than the geometric coefficient of variation.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: PK analysis set (PKS): This patient set includes all patients in the Full Analysis Set (FAS) set that have no protocol violations excluding them from PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL/mg)
Groups:
- NVP XR: Nevirapine XR (extended release)
- NVP IR: Nevirapine IR (immediate release)
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 74 | 78
(ng/mL/mg) | 15.47 (64.34) | 16.66 (75.03)
Statistical Analysis 1: Comparison: NVP XR vs NVP IR; Test type: Superiority or Other; p = 0.0080, Mixed Models Analysis; Adjusted geometric means are estimated from the mixed model for intra-individual comparison; Ratio NVP XR: NVP IR (%) = 91.20, 90% CI 2-sided [83.47 to 99.64], Standard Error of Mean 1.05

2. Secondary Outcome: AUCt,ss
Description: Area under the concentration-time curve of the Nevirapine (NVP) in plasma at steady state over the time dosing interval τ.
  All patients received nevirapine IR for 10 days prior to collection of 12-hour Area Under the Curve (AUC) data. Then, all patients were switched to nevirapine XR for 9 days prior to collection of 24-hour AUC data. The treatments of IR and XR are summarized separately using geometric means and geometric coefficients of variation.
  For NVP IR AUC measured over hours: 0,1,2,3,4,8 and 12, For NVP XR AUC measured over hours: 0,1,2,3,4,8,10,12 and 24.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: Intensive PK analysis set (IPK): This patient set includes all patients in the PK set that underwent intensive PK sampling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/ml
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
ng*h/ml
  200mg NVP XR QD (175-249 mg IR/day), n=23/22 | 99300 (37.7) | 57900 (45.7)
  300mg NVP XR QD (250-349 mg IR/day), n=11/12 | 144000 (50.1) | 58100 (35.0)
  400mg NVP XR QD (≥350 mg IR/day), n=11/15 | 108000 (60.7) | 73400 (39.8)

3. Secondary Outcome: Cmin,ss (for IR and XR Formulations by Nevirapine XR Dose Group)
Description: Minimum measured concentration of the Nevirapine in plasma at steady state over the time dosing interval τ by nevirapine XR dose group Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 21.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
ng/mL
  200 mg XR QD (175-249 mg IR/day), n=23,22 | 3090 (37.9) | 3280 (57.6)
  300 mg XR QD (250-349 mg IR/day), n=11,12 | 4160 (62.6) | 3620 (34.7)
  400 mg XR QD (≥350 mg IR/day), n=11,15 | 3410 (63.0) | 4960 (39.1)

4. Secondary Outcome: Cmax,ss (for IR and XR Formulations by Nevirapine XR Dose Group)
Description: Maximum measured concentration of the Nevirapine in plasma at steady state over the time dosing interval τ Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 22.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
ng/mL
  200 mg XR QD (175-249 mg IR/day), n=23,22 | 5350 (43.1) | 6850 (52.6)
  300 mg XR QD (250-349 mg IR/day), n=11,12 | 7970 (53.5) | 6580 (31.4)
  400 mg XR QD (≥350 mg IR/day), n=11,15 | 5890 (50.5) | 7790 (43.2)

5. Secondary Outcome: Ratio Cmax,ss/Cmin,ss
Description: Ratio of (maximum measured concentration of the Nevirapine in plasma at steady state over the time dosing interval τ)/(minimum measured concentration of the analyte in plasma at steady state over the time dosing interval τ) Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 22.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
Ratio
  200 mg XR QD (175-249 mg IR/day), n=23,22 | 1.73 (23.7) | 2.09 (32.3)
  300 mg XR QD (250-349 mg IR/day), n=11,12 | 1.91 (39.4) | 1.82 (17.8)
  400 mg XR QD (≥350 mg IR/day), n=11,15 | 1.73 (21.8) | 1.57 (21.1)

6. Secondary Outcome: %PTF
Description: Percentage peak-trough Nevirapine fluctuation, % fluctuation (degree of peak to trough fluctuation) Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 22.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
percentage fluctuation
  200 mg XR QD (175-249 mg IR/day), n=23,22 | 49.7 (47.3) | 67.9 (49.8)
  300 mg XR QD (250-349 mg IR/day), n=11,12 | 54.6 (61.1) | 59.1 (29.4)
  400 mg XR QD (≥350 mg IR/day), n=11,15 | 51.0 (47.6) | 41.5 (55.7)

7. Secondary Outcome: Tmax,ss
Description: Time from dosing to the maximum concentration of the Nevirapine in plasma at steady state over the time dosing interval τ Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 22.
  The standard deviation is actually the coefficient of variation.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
hours
  200 mg XR QD (175-249 mg IR/day), n=23,22 | 6.34 (104) [1.8 to 24.0] | 2.46 (57.9) [0.0 to 7.4]
  300 mg XR QD (250-349 mg IR/day), n=11,12 | 7.28 (121) [0.0 to 24.0] | 2.49 (50.4) [0.0 to 4.0]
  400 mg XR QD (≥350 mg IR/day), n=11,15 | 5.73 (129) [0.0 to 24.0] | 4.41 (94.2) [0.0 to 12.0]

8. Secondary Outcome: CL/F,ss
Description: Apparent clearance of the Nevirapine in the plasma after extravascular administration at steady-state Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 22.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
mL/h
  200 mg XR QD (175-249 mg IR/day), n=23,22 | 2010 (37.7) | 1780 (44.3)
  300 mg XR QD (250-349 mg IR/day), n=11,12 | 2080 (50.1) | 2240 (32.9)
  400 mg XR QD (≥350 mg IR/day), n=11,15 | 3700 (60.7) | 2640 (39.3)

9. Secondary Outcome: Cavg
Description: Average measured concentration of the Nevirapine in plasma at steady state Patients took Nevirapine (NVP) Immediate Release (IR) up to day 10 and had PK measurements taken on Day 11. This was followed by 9 days (from day 12 to day 20) taking NVP Extended Release (XR) with PK measurements taken on Day 22.
Time Frame: Day 11 prior to the next scheduled dose of Nevirapine IR and day 22 prior to the next scheduled dose of Nevirapine XR
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | NVP XR | NVP IR
Number analyzed (Participants) | 45 | 49
ng/mL
  200 mg XR QD (175-249 mg IR/day), n=23,22 | 4140 (37.7) | 4820 (45.7)
  300 mg XR QD (250-349 mg IR/day), n=11,12 | 6010 (50.1) | 4840 (35.0)
  400 mg XR QD (≥350 mg IR/day), n=11,15 | 4510 (60.7) | 6120 (39.8)

10. Secondary Outcome: Efficacy: Patients Maintaining a VL < 50 Copies/mL
Description: Patients maintaining a viral load < 50 copies/mL at Day 22.
Time Frame: Day 22
Population: Full analysis set including patients with available viral load data at day 22
Measure: Number; unit: percentage of patients
Groups:
- 3-<6 yr: Patients 3 to < 6 years old.
- 6-<12 yr: Patients 6 to < 12 years old.
- 12-<18 yr: Patients 12 to < 18 years old.
- Total.: All patients initially receive nevirapine immediate release (IR) and then all patients are switched to nevirapine extended release (XR) 100mg or 400mg tablets for a once daily dosing of 200 mg, 300 mg or 400 mg QD. After completing the PK phase patients had the option of continuing treatment with nevirapine XR in the Optional Extension Phase (OEP).
Arm/Group | 3-<6 yr | 6-<12 yr | 12-<18 yr | Total.
Number analyzed (Participants) | 25 | 23 | 31 | 79
percentage of patients | 96.0 | 100.0 | 100.0 | 98.7

11. Secondary Outcome: Efficacy: Patients Maintaining a VL < 400 Copies/mL
Description: Patients maintaining a viral load < 400 copies/mL at Day 22
Time Frame: Day 22
Population: Full analysis set including patients with available viral load data at day 22
Measure: Number; unit: percentage of patients
Arm/Group | 3-<6 yr | 6-<12 yr | 12-<18 yr | Total.
Number analyzed (Participants) | 25 | 23 | 31 | 79
percentage of patients | 100.0 | 100.0 | 100.0 | 100.0

12. Secondary Outcome: Change From Baseline in Mean CD4+ Count (Absolute)
Description: Change in mean CD4+ count (absolute) from baseline to Day 22 and from baseline to Week 24.
Time Frame: Baseline, Day 22 and week 24
Population: PK Analysis set: This patient set includes all patients in the Full Analysis Set (FAS) that have no protocol violations excluding them from PK analysis.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | 3-<6 yr | 6-<12 yr | 12-<18 yr
Number analyzed (Participants) | 24 | 24 | 31
cells/mm^3
  Day 22 | -115.6 (320.5) | 24.2 (184.8) | 60.3 (171.2)
  Week 24 (n=8;10;9) | -214.5 (397.5) | -51.2 (179.4) | 31.1 (66.4)

13. Secondary Outcome: Percentage Change From Baseline in Mean CD4+ Count
Description: ((Day 22 value-Baseline value)/Baseline value)*100. ((Week 24 value-Baseline value)/Baseline value)*100.
Time Frame: Baseline to day 22 and baseline to week 24
Population: Optional Extension Phase Treated Set (OEP TS), all patients that complete PK phase and enroll in Extension phase, and had available data at either day 22 or week 24.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 3-<6 yr | 6-<12 yr | 12-<18 yr
Number analyzed (Participants) | 24 | 24 | 31
percentage change
  Day 22 | -2.1 (6.7) | -0.0 (2.5) | 0.5 (3.6)
  Week 24 (n=8, 10, 9) | -2.1 (4.0) | -2.1 (3.4) | -1.0 (2.9)

14. Secondary Outcome: Efficacy: Patients Maintaining a VL < 50 Copies/mL at Week 24 of Optional Extension Phase
Description: Patients maintaining a viral load < 50 copies/mL at week 24 (approximately 168 days) of Optional Extension Phase (OEP).
Time Frame: week 24
Population: Full analysis set including patients with available viral load data at week 24
Measure: Number; unit: percentage of patients
Arm/Group | 3-<6 yr | 6-<12 yr | 12-<18 yr | Total.
Number analyzed (Participants) | 8 | 10 | 9 | 27
percentage of patients | 100.0 | 100.0 | 100.0 | 100.0

15. Secondary Outcome: Efficacy: Patients Maintaining a VL < 400 Copies/mL in Optional Extension Phase
Description: Patients maintaining a viral load < 400 copies/mL at week 24 of the Optional Extension Phase (OEP)
Time Frame: week 24
Population: Full analysis set including patients with available viral load data at week 24
Measure: Number; unit: percentage of patients
Arm/Group | 3-<6 yr | 6-<12 yr | 12-<18 yr | Total.
Number analyzed (Participants) | 8 | 10 | 9 | 27
percentage of patients | 100.0 | 100.0 | 100.0 | 100.0

16. Other Pre Specified Outcome: Efficacy: Patients Maintaining a VL < 50 Copies/mL at Last Available Visit
Description: Patients maintaining a viral load < 50 copies/mL at the last available visit
Time Frame: Last available visit, up to 155 weeks
Population: Optional Extension Phase Treated Set (OEP TS), all patients that complete PK phase and enroll in Extension phase with VL data available
Measure: Number; unit: percentage of patients
Arm/Group | 3-<6 yr | 6-<12 yr | 12-<18 yr | Total.
Number analyzed (Participants) | 12 | 16 | 12 | 40
percentage of patients | 100.0 | 100.0 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: From the first drug administration until 14 days after the last drug administration, up to 157 weeks
Arm/Group | Total.
Serious Adverse Events (participants affected / at risk) | 3/85
Other Adverse Events (participants affected / at risk) | 56/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total. (N=85)
Coxsackie viral infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Tonsillectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total. (N=85)
Conjunctivitis (Eye disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 8
Body tinea (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 6
Rhinitis (Infections and infestations) | 8
Tinea capitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 33
Viral upper respiratory tract infection (Infections and infestations) | 9
Headache (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 28
Rash (Skin and subcutaneous tissue disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.